CLINICAL TRIAL: NCT00362128
Title: Chinese American Cardiovascular Health Assessment CHA-CHA
Brief Title: Cardiovascular Disease Risk Factors in Chinese American Immigrants
Acronym: CHA-CHA
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Judith Wylie-Rosett, Principal Investigator, Albert Einstein College of Medicine
Other Study IDs: 2005-400; R01HL077809 (NIH)
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Hypertension; Cardiovascular Diseases; Diabetes Mellitus; Metabolic Syndrome X
Keywords: Blood Pressure, High; Obesity; Tobacco Use Disorder
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Diabetes Mellitus; Metabolic Syndrome; Obesity; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biospecimens are being analyzed to evaluate the relationship between biomarker, behaviors and sociodemographic variables. Stored specimens will permit future analysis that may involve genetic variables related to biomarker findings.
Oversight: Data Monitoring Committee: No

SUMMARY:
The Chinese population is currently the fastest growing ethnic group in New York City (NYC). Research has shown that Chinese immigrants living in NYC have higher rates of cardiovascular disease (CVD) than individuals in China. This study will evaluate the effect that acculturation has on health habits and CVD risk factors in Chinese immigrants living in NYC.

DETAILED DESCRIPTION:
CVD includes diseases that affect the heart and blood vessels. The underlying cause of CVD is atherosclerosis, in which fatty plaques develop on the inner walls of arteries. There are many risk factors for CVD, including inflammation, high blood pressure, high cholesterol, and obesity. Research has shown that CVD mortality rates differ greatly between Chinese immigrants living in NYC and individuals living in China. Because of this difference, it is important to understand the impact of immigration and acculturation on health habits and psychosocial factors, which may influence the development of CVD. This study will gather information from Chinese immigrants in NYC to identify the impact of immigration and acculturation on behavior and CVD risk factors. In addition, results from this study may provide insight into the CVD risk patterns in other immigrant groups.

This study will enroll Chinese immigrants living in NYC. Participants will attend one study visit and will complete questionnaires to assess their health habits (diet, physical activity, and smoking), stress levels, and socioeconomic status. Participants will also undergo a physical examination and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Chinese immigrant
* Currently residing in NYC

Exclusion Criteria:

* Under 18 years of age
* Not of Chinese dissent
* Born outside mainland China

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample from Chinatown region of NYC.
Sampling Method: Non-Probability Sample
Enrollment: 2072 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wylie-Rosett, EdD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- New York Downtown Hospital, New York, New York, United States

REFERENCES:
- [Derived] Lee YS, Suchday S, Wylie-Rosett J. Social support and networks: cardiovascular responses following recall on immigration stress among Chinese Americans. J Immigr Minor Health. 2015 Apr;17(2):543-52. doi: 10.1007/s10903-013-9955-9. PMID 24288021

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational: The study design was a cross-sectional observational cohort design.
Period: Overall Study
Arm/Group | Observational
Started | 2072 (Enrollment was initiated in 2007.)
Completed | 2072 (Enrollment was completed in October 2009.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Observational
Number analyzed (Participants) | 2072
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1682
  >=65 years | 390
Age, Continuous [Median (Full Range); unit: years] | 53 [21 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1093
  Male | 979
Region of Enrollment [Number; unit: participants]
  United States | 2072

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hypertension
Description: Systolic BP above 129 or Diastolic BP above 79.
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | Observational
Number analyzed (Participants) | 2072
participants | 532

ADVERSE EVENTS:
Arm/Group | Observational
Serious Adverse Events (participants affected / at risk) | 0/2072
Other Adverse Events (participants affected / at risk) | 0/2072

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No